CLINICAL TRIAL: NCT05540535
Title: Dual-Task Cost During Walking in People With Hearing Loss Compared to Normal Hearing
Brief Title: Dual-Task Cost in Bilateral Hearing Loss
Status: Completed | Type: Observational
Sponsor: New York University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY-21-01026
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2023-11

CONDITIONS: Bilateral Hearing Loss; Healthy Aging
MeSH Terms: conditions — Hearing Loss, Bilateral | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control participants with normal hearing.: Adults aged 40 and older with normal hearing will be defined as a PTA below 25dB (0.5-4 kHz) bilaterally.
  Interventions: Other: Gait assessment; Other: Cognitive assessment
- Mild Bilateral Symmetrical Hearing Loss: Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical mild HL in the past three month and on will be defined as a PTA between 26-40dB HL (0.5-4 kHz) in the better ear.
  Interventions: Other: Gait assessment; Other: Cognitive assessment
- >Moderate Bilateral Symmetrical Hearing Loss: Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical moderate, moderately-severe, severe, or profound sensorineural HL in the past three month and on.
  Moderate hearing will be defined as a PTA between 41-55dB HL (0.5-4 kHz) in the better ear, moderately-severe hearing will be defined as a PTA between 56-70dB HL (0.5-4 kHz) in the better ear, severe HL will be defined as a PTA between 71-90dB HL (0.5-4 kHz) in the better ear and profound HL will be defined as a PTA above 90+dB HL (0.5-4 kHz) in the better ear. Asymmetry of HL will be defined as a difference in PTA that is greater than dB between ears or a difference greater than/equal to 20 dB at two contiguous frequencies or greater than/equal to 10 dB at three contiguous frequencies between ears.
  Interventions: Other: Gait assessment; Other: Cognitive assessment

INTERVENTIONS:
Other: Gait assessment — The average speed of gait and spatiotemporal gait parameters would be calculated by the APDM, inertial motion units. Participants will walk in their normal speed for 1 minute along a corridor, back and forth, with or without performing a cognitive task (single or DT). The DT condition will include serial subtraction (counting backwards out loud) in jumps of 3 from a random three-digit number. Randomization of numbers will be done using the excel function generating random numbers (Excel RAND function). The numbers will be recorded for offline processing and the outcome will be the number of correct numbers. Each condition will be performed once, and all conditions will be randomized.
Other: Cognitive assessment — Participants will complete a computerized cognitive battery (CNS vital sign; CNSVS)that will include verbal memory, visual memory, Stroop test, shifting attention and 4-part continuous performance (sustained attention and working memory). Moreover, performance on the single cognitive task (serial subtraction in jumps of 3; measuring working memory and executive function) will also be evaluated while sitting (cognitive single task). The numbers will be recorded for offline processing and the outcome will be the number of correct numbers. These tests do not require the ability to hear in order to pass successfully. Also, there is a need for investigation of cognitive domains such as attention, memory, executive function, and cognitive flexibility in people with HL.

SUMMARY:
The specific aims of the research study are:

1. Compare single-task gait parameters between individuals with hearing loss (HL) and age and education matched controls with normal hearing [normal vs moderate-profound hearing loss (N=23 for each group)]. For that we will compare the primary outcome measure, gait speed, between the groups while participants are walking at a comfortable speed for 1 minute.
2. Compare cognitive function between individuals with HL and age and education matched controls. For that we will compare the Neurocognitive Index, derived from a cognitive assessment between groups.
3. Compare the effect of a cognitive task while walking on gait parameters between people with HL and age education matched controls with normal hearing. For that we will compare the primary outcome measure, gait speed, between groups while participants are walking at a comfortable speed and counting backwards [serial subtraction of 3] for 1 minute.
4. Explore whether cognitive performance (i.e., the Neurocognitive Index) is correlated with Dual task cost (DTC), a deterioration of gait speed while walking and performing concurrent cognitive task [serial subtraction of 3]. The formula to calculate this is the following: DTC = 100 X [(DT - single task)/ single task].

DETAILED DESCRIPTION:
Procedure and Data Collection:

Participants will be tested at the NYU Physical Therapy department (380 2nd Ave 3rd and 4th floors). Data will be collected by the main researcher who proposes this research work and/or two other lab researchers who are trained to conduct the full protocol. Testing will take between 1.5 to 2 hours and will always start with the cognitive assessment in order to make sure participants will perform at their best and will not be fatigued. All participants will sign an informed consent form. Participates with HL will be tested without hearing aids since recent studies suggest a possible improvement in balance as well as cognition with amplification. Participates will take off their hearing aid at the beginning of testing.

Screening Examination and Descriptive Measures of participants:

The participants will undergo a sensory systems screen including: Early Treatment Diabetic Retinopathy Study (ETDRS) chart confirming normal vision and a 5.07 monofilament screen confirming normal protective sensation at the bottom of their feet. The screening for the vestibular system will include the Dizziness Handicap Inventory (DHI) questionnaire. Screening of the auditory system will be done in participants with HL (as part of their standard care) and for healthy controls who are 60 years of age or older. Participants will also complete the following questionnaires: a demographics and anthropometrics questionnaire, and Activities-Specific Balance Confidence (ABC) to assess balance confidence. To assess the history of falls questions about past falls will be asked. The MoCA will be administered for people with normal hearing, and the HI-MoCA for people with HL in order to assess mild cognitive decline. For people with HL, the Speech, Spatial and Qualities of Hearing Scale (SSQ12), a test assessing function and interference in hearing in daily living, will be conducted. To assess balance and mobility two tests will be conducted: the modified Clinical Test of Sensory Interaction on Balance (mCTSIB) and Time Up and Go Test (TUG). First participants will wear the APDM inertial motion sensors on both feet and waist and will perform the mCTSIB. They will stand with their hands at their sides, feet together and will perform the following sensory conditions for 30 sec: (1) Stand on a firm surface with eyes open, (2) Stand on a firm surface with eyes closed, (3) Stand on a foam with eyes open, and (4) Stand on a foam with eyes closed. Secondly, participants will perform the TUG twice. The best performance in each condition out of the 2 performances will be recorded.

Cognitive Assessment:

Participants will complete a computerized cognitive battery (CNS vital sign; CNSVS) that will include verbal memory, visual memory, Stroop test, shifting attention and 4-part continuous performance (sustained attention and working memory). Moreover, performance on the single cognitive task (serial subtraction in jumps of 3; measuring working memory and executive function) will also be evaluated while sitting (cognitive single task). The numbers will be recorded for offline processing and the outcome will be the number of correct numbers. These tests do not require the ability to hear in order to pass successfully. Also, there is a need for investigation of cognitive domains such as attention, memory, executive function, and cognitive flexibility in people with HL.

Gait Assessment:

The average speed of gait and spatiotemporal gait parameters would be calculated by the APDM, inertial motion units. Participants will walk in their normal speed for 1 minute along a corridor, back and forth, with or without performing a cognitive task (single or DT). The DT condition will include serial subtraction (counting backwards out loud) in jumps of 3 from a random three-digit number. Randomization of numbers will be done using the excel function generating random numbers (Excel RAND function). The numbers will be recorded for offline processing and the outcome will be the number of correct numbers. Each condition will be performed once, and all conditions will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical moderate which is defined as a PTA between 41-55dB HL (0.5-4 kHz) in the better ear.
* Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical moderately-severe which is defined as a PTA between 56-70dB HL (0.5-4 kHz) in the better ear.
* Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical severe which is defined as a PTA between 71-90dB HL (0.5-4 kHz) in the better ear.
* Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical profound which is defined as a PTA above 90+dB HL (0.5-4 kHz) in the better ear.
* No asymmetry of HL which is defined as a difference in PTA that is greater than 15 dB between ears or a difference greater than/equal to 20 dB at two contiguous frequencies or greater than/equal to 10 dB at three contiguous frequencies between ears.
* Adults aged 40 and older with normal hearing which is defined as a PTA below 25dB (0.5-4 kHz) bilaterally.
* Subjects above 65 years of age, with symmetric ARHL in the high frequencies (>3K), with unaided PTA < 40 dB (0.5-4KHz) will be included in the control group as well.

Exclusion Criteria:

* A medical diagnosis of peripheral neuropathy.
* Lack of protective sensation based on the Semmes-Weinstein 5.07 Monofilament Test.
* Visual impairment above 20/63 (NYS Department of Motor Vehicle cutoff for driving) on the Early Treatment Diabetic Retinopathy Study (ETDRS) Acuity Test that cannot be corrected with lenses.
* Active complaint of dizziness
* Conductive HL or air bone gap
* A recent onset of a sudden HL
* Pregnancy
* Any neurological condition interfering with balance or walking (e.g. multiple sclerosis, Parkinson's disease, stroke)
* Acute musculoskeletal pain at time of testing
* Currently seeking medical care for another orthopaedic condition or vestibular rehabilitation
* Take medications that might influence gait or balance (e.g., methylphenidate);
* Inability to read an informed consent form in English.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical moderate, moderately-severe, severe, or profound sensorineural HL in the past three month and on. Normal hearing will be defined as a PTA below 25dB (0.5-4 kHz) bilaterally. Subjects above 65 years of age, with symmetric ARHL in the high frequencies (>3K), with unaided PTA < 40 dB (0.5-4KHz) will be included in the control group as well.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anat V Lubetzky, PhD, Principal Investigator — New York University
Locations (2):
- United States (2):
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - New York University Physical Therapy Department, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Control participants were recruited through the clinicaltrials.org website, the New York University community and via word of mouth. People with a clinical diagnosis of bilateral symmetrical mild, moderate, moderately-severe, severe, or profound sensorineural BHL for three months or longer were recruited from the New York Ear & Eye Institute of Mount Sinai (NYEEIMS) and the clinicaltrials.org website.
Groups:
- Control Participants With Normal Hearing.: Normal hearing will be defined as a PTA below 25dB (0.5-4 kHz) bilaterally.
- Mild Bilateral Symmetrical Hearing Loss: Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical moderate, moderately-severe, severe, or profound sensorineural HL in the past three month and on. Mild hearing will be defined as a PTA between 26-40dB HL (0.5-4 kHz) in the better ear.
Period: Overall Study
Arm/Group | Control Participants With Normal Hearing. | Mild Bilateral Symmetrical Hearing Loss | >Moderate Bilateral Symmetrical Hearing Loss
Started | 30 | 19 | 18
Completed | 28 | 16 | 15
Not Completed | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Normal Hearing: Normal hearing: according to the WHO classification43 was defined as a PTA below 25dB (0.5-4 kHz) bilaterally.
- Mild BHL: Mild BHL: according to the WHO classification43 was defined as a PTA between 25-40dB BHL(0.5-4 kHz) in the better ear.
- >Moderate BHL: Moderate BHL: according to the WHO classification43 was defined as a PTA between 41-55dB BHL(0.5-4 kHz) in the better ear.
  Moderately-severe BHL: according to the WHO classification43 was defined as a PTA between 56-70 BHL(0.5-4 kHz) in the better ear.
  Severe BHL: according to the WHO classification43 was defined as a PTA between 71-90dB BHL(0.5-4 kHz) in the better ear.
  Profound BHL: according to the WHO classification43 was defined as a PTA between 91+ dB BHL(0.5-4 kHz) in the better ear.
- Total: Total of all reporting groups
Arm/Group | Normal Hearing | Mild BHL | >Moderate BHL | Total
Number analyzed (Participants) | 28 | 16 | 15 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 2 | 5 | 24
  >=65 years | 11 | 14 | 10 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.14 (11.96) | 74.69 (8.67) | 70.93 (13.59) | 66.36 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 7 | 31
  Male | 15 | 5 | 8 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 20 | 11 | 12 | 43
  Spanish / Hispanic | 2 | 0 | 0 | 2
  Black or African American | 3 | 1 | 1 | 5
  Asian American | 2 | 2 | 0 | 4
  Asian / Pacific Islander | 0 | 1 | 0 | 1
  Alaska Native | 0 | 1 | 0 | 1
  Others | 1 | 0 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 14 | 15 | 57
  Israel | 0 | 2 | 0 | 2
Falls over the past year [Number; unit: Falls] | 5 | 5 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed (Single Task) Over 1-minute Walk
Description: The gait speed while walking for 1 min will be compared between groups. Normal gait speed will be considered 1.2-1.3 m/sec.
Time Frame: 60 seconds of a walk.
Measure: Mean (Standard Deviation); unit: m/sec
Groups:
- Mild Bilateral Symmetrical Hearing Loss: Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical Mild HL in the past three month and on.
  Mild hearing will be defined as a PTA between 26-40dB HL (0.5-4 kHz) in the better ear.
Arm/Group | Control Participants With Normal Hearing. | Mild Bilateral Symmetrical Hearing Loss | >Moderate Bilateral Symmetrical Hearing Loss
Number analyzed (Participants) | 28 | 16 | 15
m/sec | 1.14 (0.15) | 1.02 (0.21) | 1.1 (0.10)
Statistical Analysis 1: Comparison: Control Participants With Normal Hearing. vs Mild Bilateral Symmetrical Hearing Loss vs >Moderate Bilateral Symmetrical Hearing Loss; Test type: Superiority; p < 0.05, Kruskal-Wallis; The Wilcoxon signed-rank test was used for a within-group comparison

2. Primary Outcome: The Neurocognitive Index
Description: The Neurocognitive Index is the average of standardised scores obtained out of six cognitive sub-domains: Composite Memory, Reaction Time, Cognitive Flexibility, Executive Function, Working Memory and Sustained Attention, representing a form of a global score of the overall neurocognitive status of the subject. The range of the six cognitive sub-domains standardised scores and of the Neurocognitive Index is: below 70 which counts as very low score and above 110 which counts as an above averge score. Higher scores are better. Standard Scores are normalized from raw scores and present an age matched score relative to other people in a normative sample. Standardized scores have a mean of 100 and a standard deviation is 15. The schema where the mean is 100 and the standard deviation is 15 is similar to the presentation of IQ scores where the mean for normal is 100.
Time Frame: 30 minutes of assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- >Modertae Bilateral Symmetrical Hearing Loss: Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical moderate, moderately-severe, severe, or profound sensorineural HL in the past three month and on. Moderate hearing will be defined as a PTA between 41-55dB HL (0.5-4 kHz) in the better ear, moderately-severe hearing will be defined as a PTA between 56-70dB HL (0.5-4 kHz) in the better ear, severe HL will be defined as a PTA between 71-90dB HL (0.5-4 kHz) in the better ear and profound HL will be defined as a PTA above 90+dB HL (0.5-4 kHz) in the better ear. Asymmetry of HL will be defined as a difference in PTA that is greater than dB between ears or a difference greater than/equal to 20 dB at two contiguous frequencies or greater than/equal to 10 dB at three contiguous frequencies between ears.
Arm/Group | Control Participants With Normal Hearing. | Mild Bilateral Symmetrical Hearing Loss | >Modertae Bilateral Symmetrical Hearing Loss
Number analyzed (Participants) | 26 | 11 | 13
score on a scale | 105.45 (7.62) | 108.15 (5.70) | 107.05 (5.52)
Statistical Analysis 1: Comparison: Control Participants With Normal Hearing. vs Mild Bilateral Symmetrical Hearing Loss vs >Modertae Bilateral Symmetrical Hearing Loss; Test type: Superiority; p < 0.05, ANOVA

3. Primary Outcome: Gait Speed (Dual Task {DT}) Over 1-minute Walk
Description: To test allocation of attention during walking using DT paradigm the DT gait speed while walking for 1 min and performing a cognitive task which was serial subtraction (counting backwards out loud) in jumps of 3 from a random three-digit number was compared between groups.
Time Frame: 60 seconds of a walk.
Measure: Mean (Standard Deviation); unit: m/sec
Groups:
- Mild Bilateral Symmetrical Hearing Loss: Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical mild HL will be defined as a PTA between 26-40dB HL (0.5-4 kHz) in the better ear,
- > Modearte Bilateral Symmetrical Hearing Loss: Adults aged 40 and older with a clinical diagnosis of bilateral symmetrical moderate, moderately-severe, severe, or profound sensorineural HL in the past three month and on.
  Moderate hearing will be defined as a PTA between 41-55dB HL (0.5-4 kHz) in the better ear, moderately-severe hearing will be defined as a PTA between 56-70dB HL (0.5-4 kHz) in the better ear, severe HL will be defined as a PTA between 71-90dB HL (0.5-4 kHz) in the better ear and profound HL will be defined as a PTA above 90+dB HL (0.5-4 kHz) in the better ear. Asymmetry of HL will be defined as a difference in PTA that is greater than dB between ears or a difference greater than/equal to 20 dB at two contiguous frequencies or greater than/equal to 10 dB at three contiguous frequencies between ears.
Arm/Group | Control Participants With Normal Hearing. | Mild Bilateral Symmetrical Hearing Loss | > Modearte Bilateral Symmetrical Hearing Loss
Number analyzed (Participants) | 28 | 16 | 14
m/sec | 0.95 (0.20) | 0.84 (0.19) | 0.90 (0.10)
Statistical Analysis 1: Comparison: Control Participants With Normal Hearing. vs Mild Bilateral Symmetrical Hearing Loss vs > Modearte Bilateral Symmetrical Hearing Loss; Test type: Superiority; p < 0.05, Kruskal-Wallis; The Wilcoxon signed-rank test was used for a within-group comparison

4. Secondary Outcome: Single and Dual Task Stride Length
Description: Stride length while walking for one minute (single task) and while walking and counting backwards subtracting 3 from a 3 digit number (Dual task) was measures as the distance between two successive placements of the same foot. It consists of two step lengths, left and right.It was measured in meters (m).
Time Frame: 60 seconds of a walk.
Measure: Mean (Standard Deviation); unit: meter
Groups:
- Mild Bilateral Hearing Loss: Mild BHL: according to the WHO classification43 was defined as a PTA between 25-40dB BHL(0.5-4 kHz) in the better ear.
- > Moderate Bilateral Hearing Loss: Moderate BHL: according to the WHO classification43 was defined as a PTA between 41-55dB BHL(0.5-4 kHz) in the better ear.
  Moderately-severe BHL: according to the WHO classification43 was defined as a PTA between 56-70 BHL(0.5-4 kHz) in the better ear.
  Severe BHL: according to the WHO classification43 was defined as a PTA between 71-90dB BHL(0.5-4 kHz) in the better ear.
  Profound BHL: according to the WHO classification43 was defined as a PTA between 91+ dB BHL(0.5-4 kHz) in the better ear.
Arm/Group | Normal Hearing | Mild Bilateral Hearing Loss | > Moderate Bilateral Hearing Loss
Number analyzed (Participants) | 28 | 16 | 14
meter
  Single Task stride length | 1.26 (0.13) | 1.14 (0.17) | 1.20 (0.12)
  Dual Task stride length | 1.15 (0.17) | 1.02 (0.16) | 1.09 (0.13)
Statistical Analysis 1: Comparison: Normal Hearing vs Mild Bilateral Hearing Loss vs > Moderate Bilateral Hearing Loss; Test type: Superiority; p < 0.05, ANOVA

5. Secondary Outcome: Single and Dual Task Stride Time
Description: Stride time while walking for one minute (single task) and while walking and counting backwards subtracting 3 from a 3 digit number (Dual task) was measures as the time from initial contact to the next initial contact of the same foot. It was measured in seconds.
Time Frame: 60 second of a walk
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Normal Hearing | Mild BHL | >Moderate BHL
Number analyzed (Participants) | 28 | 16 | 14
seconds
  Single Task Stride time | 1.10 (0.10) | 1.14 (0.10) | 1.09 (0.06)
  Dual Task Stride time | 1.23 (0.15) | 1.24 (0.13) | 1.21 (0.12)
Statistical Analysis 1: Comparison: Normal Hearing vs Mild BHL vs >Moderate BHL; Test type: Superiority; p = 0.05, ANOVA

6. Secondary Outcome: Single and Dual Task Stride Length Variability
Description: Variability of stride length is the stride-to-stride fluctuations in walking or "gait unsteadiness"; "a measure of inconsistency and arrhythmicity of stepping". Stride Length Variability while walking for one minute (single task) and while walking and counting backwards subtracting 3 from a 3 digit number (Dual task) was measures as the coefficient of variation (CV) which is a measure of the relative variability. It was calculated as the ratio of the standard deviation to the mean. The formula to calculate that is the following: CV = 100 X (standard deviation/mean).
Time Frame: 60 second of walking
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Normal Hearing | Mild BHL | >Moderate BHL
Number analyzed (Participants) | 28 | 16 | 14
percent
  Single Task Stride Length Variability | 3.24 (1.09) | 3.60 (1.23) | 3.79 (0.84)
  Dual Task Stride Length Variability | 3.94 (1.27) | 4.96 (1.62) | 3.89 (0.95)
Statistical Analysis 1: Comparison: Normal Hearing vs Mild BHL vs >Moderate BHL; Test type: Superiority; p = 0.05, ANOVA

7. Secondary Outcome: Single and Dual Task Stride Time Variability
Description: Variability of stride time is the stride-to-stride fluctuations in walking or "gait unsteadiness"; "a measure of inconsistency and arrhythmicity of stepping". Stride Time Variability while walking for one minute (single task) and while walking and counting backwards subtracting 3 from a 3 digit number (Dual task) was measures as the coefficient of variation (CV) which is a measure of the relative variability. It was calculated as the ratio of the standard deviation to the mean. The formula to calculate that is the following: CV = 100 X (standard deviation/mean).
Time Frame: 60 second of walking
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Normal Hearing | Mild BHL | >Moderate BHL
Number analyzed (Participants) | 28 | 16 | 14
percent
  Single Task Stride Time Variability | 2.07 (0.56) | 2.37 (0.71) | 2.31 (0.62)
  Dual Task Stride Time Variability | 3.34 (1.17) | 3.59 (0.12) | 3.60 (1.33)
Statistical Analysis 1: Comparison: Normal Hearing vs Mild BHL vs >Moderate BHL; Test type: Superiority; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Through the session completion up to three hours.
Groups:
- Normal Hearing: Normal hearing: according to the WHO classification was defined as a PTA below 25dB (0.5-4 kHz) bilaterally.
- Mild BHL: Mild BHL: according to the WHO classification was defined as a PTA between 25-40dB BHL(0.5-4 kHz) in the better ear.
- > Moderate BHL: Moderate BHL: according to the WHO classification was defined as a PTA between 41-55dB BHL(0.5-4 kHz) in the better ear.
  Moderately-severe BHL: according to the WHO classification was defined as a PTA between 56-70 BHL(0.5-4 kHz) in the better ear.
  Severe BHL: according to the WHO classification was defined as a PTA between 71-90dB BHL(0.5-4 kHz) in the better ear.
  Profound BHL: according to the WHO classification was defined as a PTA between 91+ dB BHL(0.5-4 kHz) in the better ear.
Arm/Group | Normal Hearing | Mild BHL | > Moderate BHL
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/28 | 0/16 | 0/15

LIMITATIONS AND CAVEATS:
Lack of statistical power to control for covariates when splitting the BHL group to two. We ended up recruiting mostly well-treated with a high level of education, mostly exercisers and minimal comorbidities therefore findings may only be generalized to a similar demographic and to mild until moderate BHL populations. Challenges in age matching stem from difficulties recruiting young people with BHL and older adults with normal hearing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT05540535/Prot_SAP_000.pdf